CLINICAL TRIAL: NCT04144309
Title: The Effect of Acupuncture for Insomnia in Breast Cancer Patients Undergoing Chemotherapy: A Randomized, Sham-Controlled Trial
Brief Title: Acupuncture for Insomnia in Breast Cancer Patients Undergoing Chemotherapy
Acronym: BCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 19-045
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Insomnia, Secondary; Breast Cancer Female; Chemotherapy
Keywords: Acupuncture; Insomnia; Breast cancer; Chemotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True acupuncture group (Active Comparator): 12 sessions of acupuncture treatment (EA+AA) will be given twice a week for 6 weeks after randomization, followed by once a month for 3 months, for a total of 15 sessions of treatments.
  Interventions: Procedure: Electroacupuncture (EA) and Auricular Acupressure (AA)
- Sham acupuncture group (Placebo Comparator): 12 sessions of sham acupuncture treatment (SE+SA) will be given twice a week for 6 weeks after randomization, followed by once a month for 3 months, for a total of 15 sessions of treatments.
  Interventions: Procedure: Sham Electroacupuncture (SE) and Sham Auricular Acupressure (SA)

INTERVENTIONS:
Procedure: Electroacupuncture (EA) and Auricular Acupressure (AA) — EA: Ten points will be used, including GV24 (Shenting), GV20 (Baihui), EX-HN1 (Sishenchong), PC6 (Neiguan), CV12 (Zhongwan), CV4 (Guanyuan), ST25 (Tianshu), ST36 (Zusanli), SP6 (Sanyinjiao), KI3 (Taixi).
  AA: Vaccaria seeds will be embedded by acupuncturists on three auricular points (Shenmen, Sympathetic and Heart) and maintained between EA treatments.
  Arms: True acupuncture group
Procedure: Sham Electroacupuncture (SE) and Sham Auricular Acupressure (SA) — SE: The sham acupuncture treatment procedure, including the acupoint selection principle, sterilization procedure and treatment schedule, will be the same as in the acupuncture treatment group, except that sham points 1 to 2 cm exterior and inferior to the real points will be used, and no needle penetration or electric stimulation will be performed.
  SA: Three sham auricular points in the helix region (HX7, HX8, HX9) will be selected. Instead of Vaccaria seeds, soft Junci Medulla (1 to 2 mm in length, dyed black) will be used to mimic real AA with no pressure.
  Arms: Sham acupuncture group

SUMMARY:
The proposed study is a randomized, parallel-group, placebo-controlled, subject- and assessor-blind trial. It is designed according to CONSORT and STRICTA recommendations. The 138 subjects will be randomly assigned to one of the two arms using block randomization in a 1:1 ratio: (I) acupuncture treatment, and (II) sham treatment. In groups (I) and (II), acupuncture or sham acupuncture treatment will be given twice a week for 6 weeks (12 sessions). A maintenance tapering treatment schedule will then be applied once per month for 3 months (3 sessions). The primary outcome will be improvement in sleep quality as measured by the change of ISI after 6 weeks of treatment. Secondary outcome assessment tools will include PSQI, HADS, BPI, BFI, FACT-B, sleep diaries, drug diaries, blinding success questionnaire and reports of adverse events. The subjects will be scheduled for on-site follow-up assessments at 3 and 6 months after the last treatment. An intention to treat (ITT) approach will be used for data analysis.

DETAILED DESCRIPTION:
Insomnia is a frequent and disturbing symptom among cancer patients. Studies have found that cancer treatments, particularly chemotherapy, are a major cause of cancer-related insomnia. However, insomnia is under-treated in most breast cancer patients because effective, safe evidence-based treatments are lacking.

Acupuncture has been used for thousands of years to treat various diseases, including insomnia. Our previous research demonstrated the efficacy and safety of acupuncture as a treatment for insomnia. However, the effect of acupuncture on insomnia in breast cancer patients who undergo chemotherapy has been rarely studied. We propose this randomized controlled trial to examine the feasibility, effect and safety of acupuncture as a treatment for insomnia in breast cancer patients who undergo chemotherapy.

Hypothesis: We hypothesize that acupuncture is a feasible, effective and safe method for the alleviation of insomnia symptoms in breast cancer patients undergoing chemotherapy as compared with a sham control.

Primary Aim: To determine whether the insomnia condition in the acupuncture group is significantly improved when compared to the sham control group, as measured by the ISI after 6 weeks of treatment.

Secondary Aims: 1) To determine whether other sleep-related parameters in the acupuncture group improve more than those of the control group, as measured at different time points by Actiwatch, sleep diary, Pittsburgh Sleep Quality Index (PSQI), Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B), Hospital Anxiety and Depression Scale (HADS), Brief Fatigue Inventory (BFI) and Brief Pain Inventory (BPI). 2) To assess by adverse event (AE) analysis whether acupuncture is safe for treatment of insomnia in breast cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 75 years of age.
* Diagnosis of stage (American Joint Committee on Cancer (AJCC) TNM) I-IV breast cancer.
* Currently receiving chemotherapy, or have completed chemotherapy no more than 6 months.
* Insomnia onset after the diagnosis of breast cancer.
* Insomnia occurs at least 3 nights per week, and presents for at least 1 month, with fulfilment of the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnostic criteria for brief insomnia disorder Insomnia severity as defined by an ISI score of no less than 10 in the past 2 weeks.
* Expected survival time of more than 6 months.
* Ability to understand the nature of the study and willingness to give informed consent.
* Ability to provide responses during outcome measurement.

Exclusion Criteria:

* Other sleep disorder (e.g., obstructive sleep apnoea).
* Shift work or irregular sleep pattern.
* Severe visual, hearing or language defects.
* Severe hematological dysfunction (platelet count <60,000/μL, haemoglobin <8 g/dL or absolute neutrophil count <1000/μL).
* History of acupuncture use in the previous 3 months.
* Participation in other clinical trials with intervention within 3 months of the beginning of the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The primary outcome will be the change of ISI score between the baseline and the end of the 6-week treatment. The ISI is a seven-item questionnaire devised to diagnose and assess the severity of insomnia.

SECONDARY OUTCOMES:
Actiwatch | Baseline, 6 week.
  The subjects will wear Actiwatch for 1 week at baseline period and the end of 6-week treatment.
Sleep diary | Baseline, 6 week.
  Subjects will be given daily sleep diary for 1 week at baseline period and the end of 6-week treatment.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The PSQI is a reliable and valid self-reported questionnaire that assesses sleep quality over 1 month.
Hospital Anxiety and Depression Scale (HADS) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The HADS, a 14-item self-rated questionnaire, evaluates the severity of depressive and anxiety symptoms.
Brief Pain Inventory-Short Form (BPI-SF) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The BFI is a brief screening tool designed to assess the severity and impact of cancer-related fatigue on daily functioning.
Brief Fatigue Inventory (BPI) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The BPI is a self-administered questionnaire designed to assess cancer pain.
Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) | Baseline, 3 week, 6 week, 10 week, 14 week, 18 week, 30 week, 42 week.
  The FACT-B is a patient-reported outcome measure used to assess health-related quality of life in breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin ZHANG, MMed, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Hong Kong Sanatorium & Hospital, Hong Kong

REFERENCES:
- [Background] Savard J, Ivers H, Villa J, Caplette-Gingras A, Morin CM. Natural course of insomnia comorbid with cancer: an 18-month longitudinal study. J Clin Oncol. 2011 Sep 10;29(26):3580-6. doi: 10.1200/JCO.2010.33.2247. Epub 2011 Aug 8. PMID 21825267
- [Background] Savard J, Villa J, Ivers H, Simard S, Morin CM. Prevalence, natural course, and risk factors of insomnia comorbid with cancer over a 2-month period. J Clin Oncol. 2009 Nov 1;27(31):5233-9. doi: 10.1200/JCO.2008.21.6333. Epub 2009 Sep 8. PMID 19738124
- [Background] Savard J, Ivers H, Savard MH, Morin CM. Cancer treatments and their side effects are associated with aggravation of insomnia: Results of a longitudinal study. Cancer. 2015 May 15;121(10):1703-11. doi: 10.1002/cncr.29244. Epub 2015 Feb 11. PMID 25677509
- [Background] Fakih R, Rahal M, Hilal L, Hamieh L, Dany M, Karam S, Shehab L, El Saghir NS, Tfayli A, Salem Z, Assi H, Temraz S, Shamseddine A, Mukherji D. Prevalence and Severity of Sleep Disturbances among Patients with Early Breast Cancer. Indian J Palliat Care. 2018 Jan-Mar;24(1):35-38. doi: 10.4103/IJPC.IJPC_137_17. PMID 29440804
- [Background] Dahiya S, Ahluwalia MS, Walia HK. Sleep disturbances in cancer patients: underrecognized and undertreated. Cleve Clin J Med. 2013 Nov;80(11):722-32. doi: 10.3949/ccjm.80a.12170. PMID 24186891
- [Background] Cash E, Sephton SE, Chagpar AB, Spiegel D, Rebholz WN, Zimmaro LA, Tillie JM, Dhabhar FS. Circadian disruption and biomarkers of tumor progression in breast cancer patients awaiting surgery. Brain Behav Immun. 2015 Aug;48:102-14. doi: 10.1016/j.bbi.2015.02.017. Epub 2015 Feb 26. PMID 25728235
- [Background] Savard J, Morin CM. Insomnia in the context of cancer: a review of a neglected problem. J Clin Oncol. 2001 Feb 1;19(3):895-908. doi: 10.1200/JCO.2001.19.3.895. PMID 11157043
- [Background] Krystal AD. The changing perspective on chronic insomnia management. J Clin Psychiatry. 2004;65 Suppl 8:20-5. PMID 15153064
- [Background] Leung GM, Thach TQ, Lam TH, Hedley AJ, Foo W, Fielding R, Yip PS, Lau EM, Wong CM. Trends in breast cancer incidence in Hong Kong between 1973 and 1999: an age-period-cohort analysis. Br J Cancer. 2002 Oct 21;87(9):982-8. doi: 10.1038/sj.bjc.6600583. PMID 12434289
- [Background] Bergdahl L, Broman JE, Berman AH, Haglund K, von Knorring L, Markstrom A. Sleep patterns in a randomized controlled trial of auricular acupuncture and cognitive behavioral therapy for insomnia. Complement Ther Clin Pract. 2017 Aug;28:220-226. doi: 10.1016/j.ctcp.2017.06.006. Epub 2017 Jun 30. PMID 28779933
- [Background] Zia FZ, Olaku O, Bao T, Berger A, Deng G, Fan AY, Garcia MK, Herman PM, Kaptchuk TJ, Ladas EJ, Langevin HM, Lao L, Lu W, Napadow V, Niemtzow RC, Vickers AJ, Shelley Wang X, Witt CM, Mao JJ. The National Cancer Institute's Conference on Acupuncture for Symptom Management in Oncology: State of the Science, Evidence, and Research Gaps. J Natl Cancer Inst Monogr. 2017 Nov 1;2017(52):lgx005. doi: 10.1093/jncimonographs/lgx005. PMID 29140486
- [Background] Garland SN, Gehrman P, Barg FK, Xie SX, Mao JJ. CHoosing Options for Insomnia in Cancer Effectively (CHOICE): Design of a patient centered comparative effectiveness trial of acupuncture and cognitive behavior therapy for insomnia. Contemp Clin Trials. 2016 Mar;47:349-55. doi: 10.1016/j.cct.2016.02.010. Epub 2016 Mar 5. PMID 26956541
- [Background] Bao T, Goloubeva O, Pelser C, Porter N, Primrose J, Hester L, Sadowska M, Lapidus R, Medeiros M, Lao L, Dorsey SG, Badros AZ. A pilot study of acupuncture in treating bortezomib-induced peripheral neuropathy in patients with multiple myeloma. Integr Cancer Ther. 2014 Sep;13(5):396-404. doi: 10.1177/1534735414534729. Epub 2014 May 26. PMID 24867959
- [Background] Yeung WF, Chung KF, Zhang SP, Yap TG, Law AC. Electroacupuncture for primary insomnia: a randomized controlled trial. Sleep. 2009 Aug;32(8):1039-47. doi: 10.1093/sleep/32.8.1039. PMID 19725255
- [Background] Yeung WF, Chung KF, Leung YK, Zhang SP, Law AC. Traditional needle acupuncture treatment for insomnia: a systematic review of randomized controlled trials. Sleep Med. 2009 Aug;10(7):694-704. doi: 10.1016/j.sleep.2008.08.012. Epub 2009 Mar 19. PMID 19303356
- [Background] Streitberger K, Kleinhenz J. Introducing a placebo needle into acupuncture research. Lancet. 1998 Aug 1;352(9125):364-5. doi: 10.1016/S0140-6736(97)10471-8. PMID 9717924
- [Background] Zou C, Yang L, Wu Y, Su G, Chen S, Guo X, Wu X, Liu X, Lin Q. Auricular acupressure on specific points for hemodialysis patients with insomnia: a pilot randomized controlled trial. PLoS One. 2015 Apr 15;10(4):e0122724. doi: 10.1371/journal.pone.0122724. eCollection 2015. PMID 25874938
- [Background] Suen LK, Wong TK, Leung AW. Effectiveness of auricular therapy on sleep promotion in the elderly. Am J Chin Med. 2002;30(4):429-49. doi: 10.1142/S0192415X0200051X. PMID 12568272
- [Background] Savard MH, Savard J, Simard S, Ivers H. Empirical validation of the Insomnia Severity Index in cancer patients. Psychooncology. 2005 Jun;14(6):429-41. doi: 10.1002/pon.860. PMID 15376284
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Result] Yin X, Gou M, Xu J, Dong B, Yin P, Masquelin F, Wu J, Lao L, Xu S. Efficacy and safety of acupuncture treatment on primary insomnia: a randomized controlled trial. Sleep Med. 2017 Sep;37:193-200. doi: 10.1016/j.sleep.2017.02.012. Epub 2017 Mar 8. PMID 28899535
- [Derived] Mao H, Jin M, Xie L, Mao N, Shen X, Chen J, Chen X, Mao JJ, Shen X. Infrared laser moxibustion for cancer-related fatigue in breast cancer survivors: a randomized controlled trial. Breast Cancer Res. 2024 May 21;26(1):80. doi: 10.1186/s13058-024-01838-1. PMID 38773552
- [Derived] Zhang J, Qin Z, So TH, Chang TY, Yang S, Chen H, Yeung WF, Chung KF, Chan PY, Huang Y, Xu S, Chiang CY, Lao L, Zhang ZJ. Acupuncture for chemotherapy-associated insomnia in breast cancer patients: an assessor-participant blinded, randomized, sham-controlled trial. Breast Cancer Res. 2023 Apr 26;25(1):49. doi: 10.1186/s13058-023-01645-0. PMID 37101228